CLINICAL TRIAL: NCT03946475
Title: Local Specific Food-based Recommendations Developed Using Linear Programming Approach for Combating Anemia Among Adolescent Schoolgirls in Rural Indonesia
Brief Title: Remaja ASIK and Optimized Food-based Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Malang State Health Polytechnic (Unknown); Syarif Hidayatullah State Islamic University Jakarta (Other)
Responsible Party: Principal Investigator, Dr.Umi Fahmida, Principal Investigator, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RemajaASIK
Record Dates: First submitted 2019-02-23; First posted 2019-05-10 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Anemia
Keywords: Anemia; Linear programming; Optimized food based recommendations; Nutrition knowledge; Dietary intake; Dietary practices; Adolescent girls; Nutrition education; Indonesia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Intervention group (4 schools) received nutrition education in the same time. Meanwhile, control group (4 schools) did not received anything except for baseline and endline data collection.
Who Masked: Participant
Masking Description: participants did not know that they were in intervention group
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Other): 4 schools in 4 subdistrict which are divided into north and south Malang District. North area (Lawang and Singosari) and South area (Kepanjen and Gondanglegi).
  Interventions: Other: Intervention group
- Control group (No Intervention): 4 schools in 4 subdistrict which are divided into north (Sumberpucung), south (Lawang and Singosari), and east (Tumpang) Malang District.

INTERVENTIONS:
Other: Intervention group — Training of Trainers (ToT) was conducted among teacher who would deliver the messages. "Remaja ASIK" is Indonesian tagline meant "girls who are active, healthy, smart, and creative". Nutrition education was performed in every Friday, at least 30 minutes during 20 weeks. In brief, this is the key messages of optimized food based recommendations: 1) 3 meals and 2 snack every day, 2) At least 2 portions of vegetables/day including at least 5 portions/week of green leafy vegetables, 3) At least 2 portions/day of animal protein including at least 2 portions/week of liver, 4) At least 1 portion/day of tempe or tofu, 5) At least 1 portion/day of fruit, 6) At least 3 portions/week of milk.Trained teachers delivered the messages accompanied by supervisor. The delivered topics were key messages, balance nutrition, anemia, menstruation, BMI, healthy and smart, strong bone, lunch box, safe snack, and food label.
  Arms: Intervention group

SUMMARY:
Good nutritional status among adolescents is a window of opportunity to produce healthy adults or pregnant individuals. Modifying the dietary habits during adolescent girls may be a sustainable approach to ensure good nutritional status among population because those habits tend to stay for a life time. Over many years, there has much effort to overcome anemia. Iron supplementation and fortification have been the most popular and convenient strategies to combat anemia. However, there has not much success due to the high still prevalence of anemia among children and women reproductive age. Food-based approach has been defined as one of the most effective programs to combat or reduce the prevalence of anemia. In the meantime, food based recommendations (FBR) formulation through linear programming (LP) approach has been found to be more effective than the traditional method of developing FBRs called "trial and error". LP approach allows us to develop optimized diet for target population with addition to detect the nutrient problem in specific region. This study therefore aims to identify the nutrient problems in the community, to develop optimized FBR employing the LP approach and to assess effect of nutrition education using optimized FBR in order to improve the nutritional and hemoglobin status among adolescent schoolgirls in rural Malang City.

This study was conducted in several phases: 1) cross-sectional study 2) intervention study. Cross-sectional study was aimed to formulate optimized food based recommendations using linear programming. Intervention study was performed during 20 weeks with Remaja ASIK as the tagline which means Active, Healthy, Smart, and Creative. Adolescent schoolgirls aged 14-18 years was the subject of this study and 496 subjects were selected, including 152 for first phase and 344 for third phase. In addition, selected school based on inclusion criteria: 1) not boarding schools; and 2) having large number of students. In doing data collection, we collected socioecodemoghraphic data, anthropometry, biochemical data, dietary data, and cogitive performance.

DETAILED DESCRIPTION:
Nutrition among adolescent girls has been a concern in some settings throughout the world. Even in developed countries teenage girls were found to have inadequate intake of vitamins and minerals. Similarly, Indonesian adolescent girls might have suffered from similar micronutrient deficiency. Some small studies have shown that the prevalence of anemia was relatively high among adolescent girls. Over many years, there has much effort to overcome anemia. Iron supplementation and fortification have been the most popular and convenient strategies to combat anemia. However, study has shown that iron from the dietary fortification benefited the pathogens from the gut microbiota rather than increase the iron status of the host or it can cause gut inflammation among the target population.

Modifying the dietary habits during adolescent girls may be a sustainable approach to ensure good nutritional status among population because those habits tend to stay for a life time. Food-based approach has been defined as one of the most effective programs to combat or reduce the prevalence of anemia. Linear programming (LP) approach allows us to develop optimized diet for target population with addition to detect the nutrient problem in specific region. This study therefore aims to identify the nutrient problems in the community, to develop optimized food based recommendations (FBR) employing the LP approach and to assess effect of nutrition education using optimized FBR in order to improve the nutritional and hemoglobin status among adolescent schoolgirls in rural Malang City.

Eligible participants of this study were adolescent girls and meet all the inclusion criteria: 1) age: between 14-18 years 2) resident: live in rural areas of Malang district 3) willing to participate in the study 4) apparently healthy 5) already had menstruation. The list of adolescent girls from the selected high schools was obtained from each school principal. From the lists, adolescent girls was randomly selected using Random Number Apps. Those who meet the inclusion criteria was invited to participate and was given informed consent.

In the beginning of data collection, the structured interview which captures the respondents' age, address, date of birth, parents' educational and occupation, food taboo, and morbidity. The body weight was measured using SECA weighing scale and Shorr Board for height measurement. Blood specimens was collected and analyzed for levels of hemoglobin (Hb), hematocrit (Ht), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red blood cell (RBC), WBC and genetic blood disorder (hemoglobinopathy), serum ferritin, serum tranferrin receptors (TfR), and subclinincal inflammations including C-reactive protein (CRP) and a1-acid-glycoprotein (AGP). CBC analyzer was used for complete blood count whereas enzyme-linked immunoassay (ELISA) will be used to measure iron status indicators and subclinical inflammations.

Cross-sectional Study In the first phase, we conducted cross-sectional study to collect dietary data then analyzed using linear programming to obtain optimized food based recommendations. In order to develop optimized food based recommendations, we needed 152 subjects to obtain their dietary data. This sample size calculation was based on 80% power, 5% significance level, and 18.8% anemia prevalence among females and 10% absolute precision required. In the beginning of data collection, the structured interview was performed. Type of food commonly consumed and food frequency consumption per week was obtained through three days 24-hour dietary recall, 1 day weight diet record (WDR), and 3 days food records (FR). Anthropometry and biochemical measurement were assessed for each subject.

Intervention Study TIPs (Trial for Improved Practices) was conducted to pretest optimized FBR which has been developed using LP. Adolescent girls (n=20) were assessed for their actual intake using 24-hour dietary recall and last 1-week food frequency questionnaire. Afterward, they were introduced on optimized FBR and asked to practice and to write the food that are consumed in seven days food records. After one week, 24-hour dietary recall and last 1-week food frequency questionnaire were performed and group interview was conducted to identify facilitating and barriers to practicing optimized FBR.

Then, Intervention study was conducted as nutrition education in the school. As much as 144 subjects per group were randomly selected to be intervention and control group. This minimum sample size was based on 90% power, dessign effect of 2, and 20% dropout allowance. After Trial for Improved Practices (TIPs), two teachers per school were invited to join Training of Trainers (ToT) for the purpose of delivering messages of weekly nutrition education. Intervention groups received "Remaja ASIK" which is the Indonesian tagline for nutrition education in intervention schools meant "adolescent girls who are active, healthy, smart, and creative". Nutrition education was performed in every Friday, particularly in "Keputrian Session" at least 30 minutes per session during 20 weeks. Trained teachers delivered the messages of nutrition education accompanied by supervisor team. Most of materials were delivered by teaching method and several topics were delivered by poster, file presentation, showing videos and doing activities such as canteen observation, BMI calculation, and food label identification.

The effect of intervention was evaluated by nutrition knowledge, dietary intake, nutritional status, and cognitive performance. The nutrition knowledge questionnaire was generated by the team and was administered using close-ended format in baseline and endline. Dietary intake used food frequency questionnaire and three days non consecutive 24-H recall in baseline and endline. Nutritional status was determined by anthropometry and biochemical measurements. Cognitive test were administered by one well-trained enumerators who received training from psychologist to ensure standardization in the measurement and scoring procedures. Data analysis was performed using SPSS version 20. Socioeconomic status of the two groups were compared using mann-whitney test and chi-square test. The difference of changes in nutrition knowledge both of between group and within group were then analyzed by chi-square test and mcNemar test, respectively. Then, repeated measures general linear model was used to analyze the differences of dietary intake, nutritional status, and cognitive performance between group. Statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. 1st or 2nd year of high school
2. 14-18 years old
3. Apparently healthy

Exclusion Criteria:

1. Not yet menarche
2. Severe anemia (<80 g/L)
3. Having serious illness (e.g chronic kidney disease, tuberculosis)
4. Disagree to participate

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female who already had menstruation
Enrollment: 324 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (g/dL) | 20 weeks
  Hemoglobin level measured by cyanmethemoglobin in g/dL

SECONDARY OUTCOMES:
Usual iron intake (mg/day) | 20 weeks
  Measured by 3d non consecutive 24-h recalls

OTHER OUTCOMES:
Cognitive performance: attention | 20 weeks
  WISC-III Digit span measured attention. The maximum number of digits is limited to 7. Strings of digits were read by well-trained enumerators. Then, subjects were asked to re-write the number.
Cognitive performance: short-term memory | 20 weeks
  WISC-III Digit span measured short-term memory. The maximum number of digits is limited to 7. Strings of digits were read by well-trained enumerators. Then, subjects were asked to re-write the number.
Cognitive performance: processing speed | 20 weeks
  WISC-III Coding measured processing speed. In the test, symbols paired with digits are presented. Then, subjects were asked to rewrite within 120s. A score of 1 is given for each correct answer. IST captured processing speed. Well-trained enumerators asked subjects to read and to memorize given paper during 3 minutes. Then, subjects answered the questions during 6 minutes.
Cognitive performance: predictive IQ | 20 weeks
  Raven's Standard Progressive Matrices capture predictive IQ. This comprises of 5 group (10-15 questions). Subjects were asked to fill given answer sheets.
Nutrition knowledge | 20 weeks
  The nutrition knowledge questionnaire was generated by the team and was administered using close-ended format in baseline and endline data collection. The questionnaire was included 15 questions covering the following three items of nutrition knowledge: optimized food based recommendations (4 questions), anemia (4 questions), and problem nutrients and their food sources (7 questions). A positive score was corrected answer. The percentage of subjects who had corrected answer for each questions was compared between group.

CONTACTS AND LOCATIONS:
Overall Officials: Umi Fahmida, PhD, Principal Investigator — SEAMEO RECFON
Locations (1):
- Seameo Recfon, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The first co-Pi analyzed dietary intake data and the second co-Pi analyzed biomarkers data.
Supporting Information: SAP
Time Frame: 2017-now
Access Criteria: database

REFERENCES:
- [Result] Alaofe H, Zee J, Dossa R, O'Brien HT. Education and improved iron intakes for treatment of mild iron-deficiency anemia in adolescent girls in southern Benin. Food Nutr Bull. 2009 Mar;30(1):24-36. doi: 10.1177/156482650903000103. PMID 19445257
- [Result] Ferguson EL, Darmon N, Fahmida U, Fitriyanti S, Harper TB, Premachandra IM. Design of optimal food-based complementary feeding recommendations and identification of key "problem nutrients" using goal programming. J Nutr. 2006 Sep;136(9):2399-404. doi: 10.1093/jn/136.9.2399. PMID 16920861
- [Result] Fahmida U, Kolopaking R, Santika O, Sriani S, Umar J, Htet MK, Ferguson E. Effectiveness in improving knowledge, practices, and intakes of "key problem nutrients" of a complementary feeding intervention developed by using linear programming: experience in Lombok, Indonesia. Am J Clin Nutr. 2015 Mar;101(3):455-61. doi: 10.3945/ajcn.114.087775. Epub 2014 Dec 24. PMID 25733629
- [Result] Wang D, Stewart D, Chang C, Shi Y. Effect of a school-based nutrition education program on adolescents' nutrition-related knowledge, attitudes and behaviour in rural areas of China. Environ Health Prev Med. 2015 Jul;20(4):271-8. doi: 10.1007/s12199-015-0456-4. Epub 2015 Mar 15. PMID 25773683
- [Result] Blanton C. Improvements in iron status and cognitive function in young women consuming beef or non-beef lunches. Nutrients. 2013 Dec 27;6(1):90-110. doi: 10.3390/nu6010090. PMID 24379009
- [Result] Hallberg L, Hulthen L, Garby L. Iron stores and haemoglobin iron deficits in menstruating women. Calculations based on variations in iron requirements and bioavailability of dietary iron. Eur J Clin Nutr. 2000 Aug;54(8):650-7. doi: 10.1038/sj.ejcn.1601069. PMID 10951514
- [Derived] Suciyanti D, Kolopaking R, Mustafa A, Iwan S, Witjaksono F, Fahmida U. Effect of optimized food-based recommendations on nutrient intakes, hemoglobin levels, and memory performance of adolescent girls in East Java, Indonesia. Nutr J. 2025 Jan 24;24(1):13. doi: 10.1186/s12937-024-01061-w. PMID 39856679